CLINICAL TRIAL: NCT00961272
Title: An Open-Label, Pilot Study to Characterize the Pharmacokinetics of a 400mg Oral Dose of Raltegravir in the Cervicovaginal Fluids of HIV-Infected Pre-menopausal Women
Brief Title: Evaluating the Pharmacokinetics of 400 mg Oral Dose of Raltegravir in HIV-Infected Pre-Menopausal Women
Status: Completed | Type: Observational
Sponsor: Kristine Patterson, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Kristine Patterson, MD, Clinical Associate Professor of Medicine, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: 09-0889
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
Keywords: Pre-menopausal; Pharmacokinetics; Raltegravir; Women; HIV-infected
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected, pre-menopausal women

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of raltegravir in cervicovaginal fluids as compared to blood plasma of HIV-infected pre-menopausal women.

DETAILED DESCRIPTION:
Participants: Six HIV-positive pre-menopausal women already undergoing therapy with raltegravir.

Procedures (methods): This study will be conducted at a single site: the University of North Carolina at Chapel Hill. An outpatient screening visit will assess subject suitability and willingness to participate. During one pharmacokinetic visit women will be asked to self-collect cervicovaginal samples using a cervicovaginal fluid aspirator at the following time points: pre-dose and 1, 2, 4, 6, 8, 10, and 12 hours after raltegravir 400mg dose administration. One 3mL EDTA tube will be collected at the same time points to analyze blood plasma. A follow-up safety visit will be completed within 30 days of the inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by HIV serology or detectable viral load
* Able to provide informed consent
* In the opinion of the investigator, able to comply with their treatment regimen and study procedures
* Currently receiving raltegravir as treatment for HIV infection. Subjects must have been on raltegravir for at least 3 weeks prior to the inpatient pharmacokinetic sampling stay.
* All women of reproductive potential (who have not reached menopause or undergone bilateral oophorectomy, or tubal ligation) must have a negative serum β-HCG pregnancy test performed at screening.
* Subjects must test negative for sexually transmitted infections (gonorrhea, chlamydia, trichomonas, bacterial vaginosis, or syphilis) at screening
* All study volunteers must agree not to participate in a conception process (e.g., active attempt to become pregnant).
* Subjects must be willing to abstain from intercourse, and vaginal instrumentation, including douching, within the 48 hours prior to all study visits.
* If participating in sexual activity that could lead to pregnancy between study visits, the female study volunteer/male partner must use at least one reliable method of contraception (e.g., condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD)

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Any condition which in the opinion of the investigator is likely to interfere with follow-up or ability to take the study medication appropriately
* A positive test for bacterial vaginosis, syphilis, gonorrhea, chlamydia, or trichomonas

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Six HIV-infected adult pre-menopausal women (> or equal to 18 and less than or equal to 49 years of age) currently undergoing treatment with raltegravir with an intact uterus and cervix will be considered for enrollment. Pregnant women and women testing positive for STDs (bacterial vaginosis, syphilis, gonorrhea, chlamydia, or trichomonas) will be excluded. The six HIV-infected women enrolled in this study will come from the UNC-Chapel Hill Infectious Diseases Clinic and associated clinics in local Health Departments.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To describe the pharmacokinetics of raltegravir in cervicovaginal secretions as compared to blood plasma at steady-state in six HIV-positive women. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Patterson, MD, Principal Investigator — University of North Carolina, Chapel Hill; Angela Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Musicco M, Lazzarin A, Nicolosi A, Gasparini M, Costigliola P, Arici C, Saracco A. Antiretroviral treatment of men infected with human immunodeficiency virus type 1 reduces the incidence of heterosexual transmission. Italian Study Group on HIV Heterosexual Transmission. Arch Intern Med. 1994 Sep 12;154(17):1971-6. PMID 8074601
- [Background] Otten RA, Smith DK, Adams DR, Pullium JK, Jackson E, Kim CN, Jaffe H, Janssen R, Butera S, Folks TM. Efficacy of postexposure prophylaxis after intravaginal exposure of pig-tailed macaques to a human-derived retrovirus (human immunodeficiency virus type 2). J Virol. 2000 Oct;74(20):9771-5. doi: 10.1128/jvi.74.20.9771-9775.2000. PMID 11000253
- [Background] Lallemant M, Jourdain G, Le Coeur S, Mary JY, Ngo-Giang-Huong N, Koetsawang S, Kanshana S, McIntosh K, Thaineua V; Perinatal HIV Prevention Trial (Thailand) Investigators. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med. 2004 Jul 15;351(3):217-28. doi: 10.1056/NEJMoa033500. Epub 2004 Jul 9. PMID 15247338
- [Background] Blankson JN, Persaud D, Siliciano RF. The challenge of viral reservoirs in HIV-1 infection. Annu Rev Med. 2002;53:557-93. doi: 10.1146/annurev.med.53.082901.104024. PMID 11818490
- [Background] Pierson T, Hoffman TL, Blankson J, Finzi D, Chadwick K, Margolick JB, Buck C, Siliciano JD, Doms RW, Siliciano RF. Characterization of chemokine receptor utilization of viruses in the latent reservoir for human immunodeficiency virus type 1. J Virol. 2000 Sep;74(17):7824-33. doi: 10.1128/jvi.74.17.7824-7833.2000. PMID 10933689
- [Background] Markowitz M, Morales-Ramirez JO, Nguyen BY, Kovacs CM, Steigbigel RT, Cooper DA, Liporace R, Schwartz R, Isaacs R, Gilde LR, Wenning L, Zhao J, Teppler H. Antiretroviral activity, pharmacokinetics, and tolerability of MK-0518, a novel inhibitor of HIV-1 integrase, dosed as monotherapy for 10 days in treatment-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):509-15. doi: 10.1097/QAI.0b013e31802b4956. PMID 17133211
- [Background] Cohen MS. Preventing sexual transmission of HIV. Clin Infect Dis. 2007 Dec 15;45 Suppl 4:S287-92. doi: 10.1086/522552. PMID 18190301
- [Background] Isentress (raltegravir) Prescribing Guide. Merck & Co, Inc. October 2007